CLINICAL TRIAL: NCT00132093
Title: The Effects of Eplerenone on Left Ventricular Remodelling Post-Acute Myocardial Infarction: a Double-Blind Placebo-Controlled Cardiac MR-Based Study
Brief Title: Effects of Eplerenone on Left Ventricular Remodelling Following Heart Attack
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WN04CA024; Eudract number 2004-004399-35
Record Dates: First submitted 2005-08-18; First posted 2005-08-19 (Estimated); Last update posted 2006-04-10 (Estimated); Status verified 2004-11

CONDITIONS: Myocardial Infarction
Keywords: Left ventricular remodelling; Acute myocardial infarction; Left ventricular dysfunction; Eplerenone; Cardiac Magnetic Resonance Imaging
MeSH Terms: conditions — Myocardial Infarction; Ventricular Dysfunction, Left | interventions — Eplerenone

INTERVENTIONS:
Drug: Eplerenone

SUMMARY:
The purpose of this study is to ascertain whether treatment with the drug eplerenone, taken early after a heart attack, prevents or reduces some of the adverse changes that may otherwise naturally occur within the heart muscle, that lead ultimately to weakening of the heart muscle and premature death.

DETAILED DESCRIPTION:
Despite advances in detection and treatment of coronary artery disease, and numerous campaigns to promote healthier lifestyles, ischaemic heart disease (IHD) remains very common worldwide but particularly in the West of Scotland. Following a heart attack, the main pumping chamber - the left ventricle (LV) - will be significantly damaged in around 40% of patients to the extent that it fails to pump as effectively as before. Despite current medical treatment, this failing LV slowly but continuously deteriorates with time (this is known as LV remodelling), which can lead to "heart failure".

Eplerenone, a hormone blocker (aldosterone antagonist), has been shown to reduce death rates and improve symptoms in patients with acute heart attacks - or myocardial infarctions (MI)- who additionally have impaired LV function and heart failure (or diabetes). The researchers assume that eplerenone may exert some of these beneficial effects by preventing or reducing this LV remodelling process.

Cardiac MRI provides very accurate assessment of LV function, such that small numbers of patients only are required to detect differences in LV function over time when comparing one group against another. The researchers are therefore comparing sequential cardiac MRI appearances and measurements in patients with acute MI and LV impairment at baseline (within 2 weeks of the acute MI), 3 months and 6 months. After the first MRI scan, patients are assigned to eplerenone or placebo in addition to usual secondary preventive therapy (double-blinded), which continues for 6 months, after which each patient's involvement in the trial is finished.

As eplerenone has been shown to benefit those with acute MI plus LV impairment and heart failure (or diabetes), such patients cannot ethically be put into a trial in which they may potentially be placed in a placebo group. For this reason, a slightly different cohort of patients are being used - acute MI with LV impairment but without clinical heart failure or diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or above
2. Acute myocardial infarction within last 1-14 days (defined by typical electrocardiogram [ECG] changes and/or elevated cardiac enzymes to at least twice the upper limit of normal)
3. Left ventricular systolic dysfunction (LVSD) based on echocardiographic wall motion score index (WMSI) and left ventricular ejection fraction (LVEF) < 40%
4. Ability to give written informed consent

Exclusion Criteria:

1. Clinical or radiological heart failure
2. Established diabetes mellitus
3. Current use of potassium (K)-sparing diuretics, clarithromycin, nefazodone, itraconazole, ketoconazole, ritonavir, nelfinavir, tacrolimus, cyclosporin.
4. Serum creatinine > 220 µmol/l
5. Serum potassium > 5.0 mmol/l
6. Pregnancy
7. Addison's disease
8. MRI-incompatible (ferrous) sulphate prosthesis
9. Claustrophobia (unable to tolerate MR environment)
10. Concurrent use of phenytoin, carbamazepine, rifampicin or St. John's Wort (reduce efficacy of eplerenone).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-04

PRIMARY OUTCOMES:
Change in left ventricular (LV) end-systolic volume over 6 months, based on cardiac magnetic resonance imaging (MRI) measurements, comparing treatment group to placebo group

SECONDARY OUTCOMES:
Comparison of lab blood markers of LV remodelling over 6 months, comparing treatment group to placebo group
Comparison of neurohormonal levels over 6 months, comparing treatment group to placebo group
Comparison of cardiac electrical stability (heart rate variability, QT dispersion) over 6 months, comparing treatment group to placebo group
Analysis of DNA at baseline between and within the eplerenone group and the control group - to see if mutations in the gene that encodes aldosterone synthase - CYP112B - predict remodelling and response to aldosterone blockade

CONTACTS AND LOCATIONS:
Overall Officials: Robin AP Weir, MBChB, BSc, MRCP, Principal Investigator — NHS Greater Glasgow and Clyde; Henry J Dargie, MBChB,FRCP, Study Director — NHS Greater Glasgow and Clyde; John JV McMurray, FRCP,MD,FESC, Study Director — University of Glasgow
Locations (1):
- Western Infirmary, Glasgow, Scotland, United Kingdom

REFERENCES:
- [Background] Pitt B, Remme W, Zannad F, Neaton J, Martinez F, Roniker B, Bittman R, Hurley S, Kleiman J, Gatlin M; Eplerenone Post-Acute Myocardial Infarction Heart Failure Efficacy and Survival Study Investigators. Eplerenone, a selective aldosterone blocker, in patients with left ventricular dysfunction after myocardial infarction. N Engl J Med. 2003 Apr 3;348(14):1309-21. doi: 10.1056/NEJMoa030207. Epub 2003 Mar 31. PMID 12668699
- [Derived] Weir RA, Petrie CJ, Murphy CA, Clements S, Steedman T, Miller AM, McInnes IB, Squire IB, Ng LL, Dargie HJ, McMurray JJ. Galectin-3 and cardiac function in survivors of acute myocardial infarction. Circ Heart Fail. 2013 May;6(3):492-8. doi: 10.1161/CIRCHEARTFAILURE.112.000146. Epub 2013 Mar 15. PMID 23505301
- [Derived] Weir RA, Tsorlalis IK, Steedman T, Dargie HJ, Fraser R, McMurray JJ, Connell JM. Aldosterone and cortisol predict medium-term left ventricular remodelling following myocardial infarction. Eur J Heart Fail. 2011 Dec;13(12):1305-13. doi: 10.1093/eurjhf/hfr129. Epub 2011 Sep 22. PMID 21940729
- [Derived] Weir RA, Clements S, Steedman T, Dargie HJ, McMurray JJ, Squire IB, Ng LL. Plasma TIMP-4 predicts left ventricular remodeling after acute myocardial infarction. J Card Fail. 2011 Jun;17(6):465-71. doi: 10.1016/j.cardfail.2011.02.002. Epub 2011 Mar 25. PMID 21624734
- [Derived] Weir RA, Murphy CA, Petrie CJ, Martin TN, Balmain S, Clements S, Steedman T, Wagner GS, Dargie HJ, McMurray JJ. Microvascular obstruction remains a portent of adverse remodeling in optimally treated patients with left ventricular systolic dysfunction after acute myocardial infarction. Circ Cardiovasc Imaging. 2010 Jul;3(4):360-7. doi: 10.1161/CIRCIMAGING.109.897439. Epub 2010 Mar 26. PMID 20348438
- [Derived] Weir RA, Miller AM, Murphy GE, Clements S, Steedman T, Connell JM, McInnes IB, Dargie HJ, McMurray JJ. Serum soluble ST2: a potential novel mediator in left ventricular and infarct remodeling after acute myocardial infarction. J Am Coll Cardiol. 2010 Jan 19;55(3):243-50. doi: 10.1016/j.jacc.2009.08.047. PMID 20117403
- [Derived] Weir RA, Martin TN, Murphy CA, Petrie CJ, Clements S, Steedman T, Dargie HJ, Wagner GS. Comparison of serial measurements of infarct size and left ventricular ejection fraction by contrast-enhanced cardiac magnetic resonance imaging and electrocardiographic QRS scoring in reperfused anterior ST-elevation myocardial infarction. J Electrocardiol. 2010 May-Jun;43(3):230-6. doi: 10.1016/j.jelectrocard.2010.01.003. Epub 2010 Feb 1. PMID 20116803
- [Derived] Weir RA, Mark PB, Petrie CJ, Clements S, Steedman T, Ford I, Ng LL, Squire IB, Wagner GS, McMurray JJ, Dargie HJ. Left ventricular remodeling after acute myocardial infarction: does eplerenone have an effect? Am Heart J. 2009 Jun;157(6):1088-96. doi: 10.1016/j.ahj.2009.04.001. PMID 19464421
- [Derived] Iraqi W, Rossignol P, Angioi M, Fay R, Nuee J, Ketelslegers JM, Vincent J, Pitt B, Zannad F. Extracellular cardiac matrix biomarkers in patients with acute myocardial infarction complicated by left ventricular dysfunction and heart failure: insights from the Eplerenone Post-Acute Myocardial Infarction Heart Failure Efficacy and Survival Study (EPHESUS) study. Circulation. 2009 May 12;119(18):2471-9. doi: 10.1161/CIRCULATIONAHA.108.809194. Epub 2009 Apr 27. PMID 19398668
- [Derived] Weir RA, Chong KS, Dalzell JR, Petrie CJ, Murphy CA, Steedman T, Mark PB, McDonagh TA, Dargie HJ, McMurray JJ. Plasma apelin concentration is depressed following acute myocardial infarction in man. Eur J Heart Fail. 2009 Jun;11(6):551-8. doi: 10.1093/eurjhf/hfp043. Epub 2009 Apr 6. PMID 19351633
- [Derived] Weir RA, Martin TN, Petrie CJ, Murphy A, Clements S, Steedman T, Wagner GS, McMurray JJ, Dargie HJ. Cardiac and extracardiac abnormalities detected by cardiac magnetic resonance in a post-myocardial infarction cohort. Cardiology. 2009;113(1):1-8. doi: 10.1159/000161233. Epub 2008 Oct 10. PMID 18849604